CLINICAL TRIAL: NCT02542514
Title: Phase II Study of Ibrutinib in Patients With Relapsed or Refractory Primary Central Nervous Lymphoma or Intraocular Lymphoma
Brief Title: Study of Ibrutinib in Patients With Relapsed or Refractory Primary Central Nervous Lymphoma or Intraocular Lymphoma
Acronym: iLOC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iLOC
Record Dates: First submitted 2015-08-31; First posted 2015-09-07 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Primary Central Nervous Lymphoma; Intraocular Lymphoma
Keywords: PCNSL; IOL
MeSH Terms: conditions — Intraocular Lymphoma | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ibrutinib (Experimental): ibrutinib in monotherapy 28 days/cycles
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — p.o. 560 mg once a day (four 140 mg capsules) for one year (12 cycles of 28 days)

SUMMARY:
The study is an open label, prospective, multicenter, phase II study which aims to define ibrutinib efficacy in patients with relapsed or refractory primary central nervous lymphoma (PCNSL) or intraocular lymphoma (IOL) as measured by the disease control (DC) rate (complete response (CR) + uncertain complete response (Ru) + partial response (PR) stabilized disease (SD)) after 2 cycles of treatment according to International study group for PCNSL (IPCG) criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of PCNSL or cytologically proven diagnosis of IOL or lymphomatous meningitis of B-cell type. In case of CNS lymphoma relapse or refractory PCNSL, cerebral biopsies are not required if imaging reveals typical images of PCNSL. In case of isolated IOL relapse, vitrectomy is not required if i) vitrectomy was part of the initial diagnosis workout, and ii) ocular examination and dosage of IL-10 in the anterior chamber of the eye performed at relapse or progression are highly in favour of IOL relapse (> 50 pg/ml in aqueous humor or 400 pg/ml in vitreous).
2. Aged 18 years and older.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2.
4. Life expectancy ≥ 3 months.
5. No more than 4 lines of anti-cancer treatment received.
6. Patients must have recovered within 28 days to a grade ≤ 1 from all toxicities related to prior treatments.
7. Adequate Laboratory Parameters within 14 days:
8. Measurable PCNSL as diagnosed on MRI
9. Highly effective method of birth control during and after the study consistent. Men must agree to not donate sperm during and after the study. These restrictions apply for 1 year after the last dose of study drug.
10. Women of childbearing potential must have a negative serum beta-hCG or urine pregnancy test at Screening.
11. Sign of an informed consent document.The informed consent document can be signed by a person of confidence in case neurologic disorders related to the disease prevent the patient to sign himself.

Exclusion Criteria:

1. Contraindication to any excipients of the drug.
2. T-cell lymphoma.
3. Prior history of malignancies other than lymphoma (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast), prior history of systemic lymphoma, unless the patient has been free of the disease for ≥ 3 years.
4. Prior history of organ transplantation or other cause of severe immunodeficiency.
5. Major surgery, within 4 weeks prior to the first dose of study drug.
6. History of stroke or intracranial hemorrhage within 6 months prior to randomization. Patients with post-biopsies hemorrhagic sequela defined as a small hyperdense lesion < 3 mm on T2* sequence won't be excluded.
7. Requires anticoagulation with warfarin or equivalent vitamin K antagonists or ongoing warfarin medication or other equivalent vitamin K antagonists.
8. Any anti-platelet aggregant medication except acetyl salicylic acid ≤ 75 mg/day.
9. Requires treatment with strong CYP3A4 inhibitors.
10. Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 or Class 4 cardiac disease as defined by the New York Heart Association Functional Classification.
11. Vaccinated with live, attenuated vaccines within 4 weeks prior to the first dose of study drug.
12. Known history of HIV or active Hepatitis C Virus (HCV; RNA polymerase chain reaction [PCR]-positive) or active Hepatitis B Virus (HBs Ag positive or DNA PCR-positive) infection or any uncontrolled active systemic infection requiring intravenous (IV) antibiotics.
13. Any life-threatening illness, medical condition, or organ system dysfunction which could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk.
14. Inability to swallow capsules.
15. Pregnancy or lactation.
16. Use of anti-cancer drug therapy within 21 days prior to the first dose of study drug.
17. Previous treatment by BTK inhibitors and PI3K inhibitors.
18. Known bleeding diathesis.
19. Inclusion in another experimental anti-cancer drug therapy*.
20. Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.
21. Patient under measure of legal protection.
22. No social security affiliation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
disease control rate (CR + CRu + PR +SD) | 2 months
  Disease control (DC) rate (CR + CRu + PR + SD) after 2 cycles of treatment according to IPCG criteria.

SECONDARY OUTCOMES:
Number of AE | 12 months
  To evaluate tolerance and toxicity of ibrutinib.
disease control | 4, 6, 9 and 12 months
  according to IPCG criteria evaluated locally by investigators and the results of the MRI review (maximum of 6 MRI review per patient).
overall response (OR) | 4, 6, 9 and 12 months
  according to IPCG criteria evaluated locally by investigators and the results of the MRI review (maximum of 6 MRI review per patient).
complete response (CR) rate | 4, 6, 9 and 12 months
  according to IPCG criteria evaluated locally by investigators and the results of the MRI review (maximum of 6 MRI review per patient).
overall survival (OS) | 4, 6, 9 and 12 months
  according to IPCG criteria evaluated locally by investigators and the results of the MRI review (maximum of 6 MRI review per patient).
time to progression | 12 months
progression-free survival (PFS) | 12 months

OTHER OUTCOMES:
concentration of ibrutinib in cerebrospinal fluid | baseline and 2 months
  Pharmacokinetics of ibritunib in the cerebrospinal fluid.

CONTACTS AND LOCATIONS:
Overall Officials: Carole Soussain, MD, Study Chair — Lymphoma Study Association
Locations (10):
- France (10):
  - CHU d'ESTAING, Clermont-Ferrand
  - CHU de Grenoble, Grenoble
  - CHRU de LILLE - Claude Huriez, Lille
  - Centre Léon Bérard, Lyon
  - CHU de la Pitié Salpêtrière, Paris
  - CHU de la Timone, Paris
  - CHU de Rennes, Rennes
  - Centre Henri Becquerel, Rouen
  - Hôpital René Huguenin Institut Curie, Saint-Cloud
  - CHU Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Soussain C, Choquet S, Blonski M, Leclercq D, Houillier C, Rezai K, Bijou F, Houot R, Boyle E, Gressin R, Nicolas-Virelizier E, Barrie M, Molucon-Chabrot C, Lelez ML, Clavert A, Coisy S, Leruez S, Touitou V, Cassoux N, Daniau M, Ertault de la Bretonniere M, El Yamani A, Ghesquieres H, Hoang-Xuan K. Ibrutinib monotherapy for relapse or refractory primary CNS lymphoma and primary vitreoretinal lymphoma: Final analysis of the phase II 'proof-of-concept' iLOC study by the Lymphoma study association (LYSA) and the French oculo-cerebral lymphoma (LOC) network. Eur J Cancer. 2019 Aug;117:121-130. doi: 10.1016/j.ejca.2019.05.024. Epub 2019 Jul 3. PMID 31279304